CLINICAL TRIAL: NCT02597647
Title: Bacterial Composition and Immune Responses in the Nose and Oropharynx During Influenza Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: J. Craig Venter Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#11-000326-CR-00003
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Influenza
Keywords: immunology; Microbiota
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Live attenuated influenza vaccine (Experimental): Healthy adult volunteers given intranasal FluMist (Live Attenuated Influenza vaccine). Subjects will undergo nasal swabs, nasopharyngeal washes, and nasal epithelial brushings at baseline, 1-2 weeks, and 4-6 weeks after LAIV.
  Interventions: Biological: LAIV
- Saline nasal spray (Placebo Comparator): Healthy adult volunteers given intranasal saline nasal spray. Subjects will undergo nasal swabs, nasopharyngeal washes, and nasal epithelial brushings at baseline, 1-2 weeks, and 4-6 weeks after saline administration.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: LAIV — Subjects underwent nasal swabs, nasopharyngeal saline wash, and nasal brushings pre, and 1-2 weeks and 4-6 weeks following intranasal administration of LAIV.
  Arms: Live attenuated influenza vaccine
Other: Saline — Subjects underwent nasal swabs, nasopharyngeal saline wash, and nasal brushings pre, and 1-2 weeks and 4-6 weeks following intranasal administration of saline nasal spray.
  Other Names: Ocean spray
  Arms: Saline nasal spray

SUMMARY:
This study will serve to determine how influenza infection alters the bacterial colonization patterns in the nasal and oropharyngeal compartments, and whether the immune response correlate with these alterations. The investigators will be determining bacterial composition and immune responses in the nose and oropharynx during influenza infection.

Specific Aims

Therefore, the overall aims of this study are as follows:

1. To identify baseline composition and kinetic changes in the nasal and oropharyngeal microflora and immune responses after administering intranasal live attenuated influenza virus (i.e., FluMist® vaccine) or saline mist to healthy subjects;
2. To identify nasal and oropharyngeal microbial composition and local immune responses during influenza infections and after resolution of infection, and correlate these changes with clinical outcomes.

DETAILED DESCRIPTION:
Randomization and Post-Randomization Visits After undergoing the nasal swabs and nasopharyngeal washes, and nasal epithelial brushing, healthy volunteers will be randomly assigned to receive either saline nasal spray (placebo) or FluMist® nasal influenza vaccine (live attenuated influenza vaccine, or LAIV). They will return 1-2 weeks and 4-6 weeks later to repeat the nasal swabs and nasopharyngeal washes, and nasal epithelial brushings done at the Enrollment Visit.

Samples will be processed to isolate 16s bacterial RNA and host RNA. 16s rRNA will be analyzed by 16S sequencing for to determine the composition of the bacterial microbiome pre and post LAIV or saline (placebo) administration. Host immune responses will be assessed based upon microarray analysis of host RNA pre and post LAIV or saline administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:
* Healthy subjects between the ages of 18 and 65. Approximately half of the subjects will be female and approximately half will be male.
* Must be eligible to receive live-attenuated nasal version of the influenza vaccine.
* Must be able to provide signed and dated informed consent.
* Healthy subjects willing and able to provide oropharyngeal and nasal cavity specimens

Exclusion Criteria:

* Immunosuppressive conditions or medications
* chronic systemic medical illness
* infections or antibiotic use within the past 60 days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changes in the bacterial composition (Bacterial "microbiome") over time | Changes from baseline at 1-2 weeks and 4-6 weeks after LAIV or saline spray
  isolation of 16S RNA from nasal swabs and nasopharyngeal washes for 16S sequencing for bacterial microbiome
Changes in gene expression in the nasal lining of study participants | Changes from baseline at 1-2 weeks after LAIV or saline spray
  RNA isolation from nasal brushes which will undergo microarray analysis to measure changes in immune gene expression

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Tarabichi Y, Li K, Hu S, Nguyen C, Wang X, Elashoff D, Saira K, Frank B, Bihan M, Ghedin E, Methe BA, Deng JC. The administration of intranasal live attenuated influenza vaccine induces changes in the nasal microbiota and nasal epithelium gene expression profiles. Microbiome. 2015 Dec 15;3:74. doi: 10.1186/s40168-015-0133-2. PMID 26667497